CLINICAL TRIAL: NCT06785519
Title: A Clinical Study of the Safety and Efficacy of CD19/BCMA CAR-T Cell Therapy for Refractory/Relapsed Lupus Nephritis
Brief Title: CD19/BCMA CAR-T Cell Therapy for Refractory/Relapsed Lupus Nephritis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: He Huang (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Sponsor-Investigator, He Huang, Clinical Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024012
Record Dates: First submitted 2025-01-13; First posted 2025-01-21 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-10

CONDITIONS: Lupus Nephritis
Keywords: CD19/BCMA CAR-T
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lupus Nephritis (Experimental): Administration of CD19/BCMA Lupus Nephritis Targeted CAR T-cells
  Interventions: Biological: CD19/BCMA Lupus Nephritis Targeted CAR T-cells injection

INTERVENTIONS:
Biological: CD19/BCMA Lupus Nephritis Targeted CAR T-cells injection — Each subject receive CD19/BCMA Lupus Nephritis Targeted CAR T-cells by intravenous infusion

SUMMARY:
A Clinical Study of the Safety and Efficacy of CD19/BCMA CAR-T Cell Therapy for Refractory/Relapsed Lupus Nephritis.

DETAILED DESCRIPTION:
In this study, 9 patients with relapsed refractory Lupus Nephritis were proposed to undergo CD19/BCMA CAR-T Cells therapy. Under the premise that its safety has been clarified in previous studies, further observation and evaluation of the effectiveness of CD19/BCMA CAR-T Cells therapy for relapsed refractory Lupus Nephritis; At the same time, on the basis of expanding the sample size, more safety data on CD19/BCMA CAR-T Cells treatment for relapsed refractory Lupus Nephritis were accumulated.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old;
* 2. A clinical diagnosis of systemic lupus erythematosus (SLE) according to the 2019 American College of Rheumatology (ACR) and European Federation of Rheumatology Societies (EULAR) /ACR classification criteria. Grade III, IV, or V lupus nephritis was confirmed by biopsy according to the 2003 ISN/RPS standard.
* 3. SLEDAI-2K ≥8 during screening
* 4. failure to respond to two or more standard immunosuppressive therapies, or relapse (increased disease activity index and need to adjust drug dose or type);
* 5. Expected survival >12 weeks;
* 6. Fertile women and men agree to use appropriate contraceptive methods before entering the study, during study participation, and for 6 months after transfusion (the safety of this therapy for the unborn child is not known);
* 7. Volunteer to participate in this experiment and sign the informed consent.

Exclusion Criteria:

* 1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular hemorrhagic diseases;
* 2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
* 3. Active infected persons who are not cured:
* 4. Active hepatitis B or C virus infection;
* 5. Patients who have taken more than 20mg/d of prednisone or equivalent systemic steroid drugs within 1 week prior to treatment (except those who have recently or currently taken inhaled steroids);
* 6. Have used any gene therapy products before;
* 7. Insufficient amplification ability (<5 times) in response to CD3 / CD28 costimulation signals;
* 8. ALT/AST>3 times the normal amount or bilirubin >2.0 mg/dl;
* 9. Those who have other uncontrolled diseases that the researcher deems unsuitable for enrollment;
* 10. HIV-infected people;
* 11. Any situation that the investigator believes may increase the risk to the subject or interfere with the test results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-01-31 (Estimated); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 years after Treatment
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Urinary protein index | Up to 24 hours after Treatment
  Urinary protein index（24h urinary protein、Urinary protein/creatinine ratio）

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China